CLINICAL TRIAL: NCT02572011
Title: A Games-console Based Balance Training Intervention for Transtibial Amputees: A Randomised Controlled Trial
Brief Title: Transtibial Amputee Balance Training: A Randomised Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Nottingham Trent University (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University of Hull (Other); Bournemouth University (Other); Jonkoping University (Other)
Responsible Party: Principal Investigator, Dr. Cleveland T. Barnett, Senior Lecturer in Biomechanics, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NTU127818
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Lower Limb Amputation
Keywords: Lower limb amputation; Transtibial; Balance; Postural Control; Limits of Stability; Rehabilitation; Home-based intervention; Nintendo Wii; Balance Board

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants in the control (CON) group will not complete any formalised balance training as part of the current study.
- Experimental (Experimental): Participants in the experimental group will complete the Home-based Games Console Balance Training intervention.
  Interventions: Other: Home-based Games Console Balance Training

INTERVENTIONS:
Other: Home-based Games Console Balance Training — The balance training intervention involves completing prescribed balance tasks for a minimum of 60 minutes per session, three times a week for 12 weeks (minimum intervention time of 2160 minutes) in their own home. Participants will perform the balance related Wii Fit games that have been suggested previously by professional bodies and amputee therapists (BACPAR Ossur Wii Fit Exercise Recommendations).
  Arms: Experimental

SUMMARY:
Lower limb amputees have reduced joint mobility and strength which negatively influence an individual's ability to maintain balance. Individuals with lower limb amputation also have an increased fear of falling and reduced social participation because of this fear. Improving balance ability, reducing falls and fear of falling through effective balance training interventions would have a number of socio-economic benefits. The aim of the current study is to investigate whether taking part in a games console based-balance intervention, improves balance ability in individuals with lower limb amputation.

DETAILED DESCRIPTION:
Lower limb amputation (LLA) results in the loss of the biological joint structures such as the ankle and knee, along with the associated musculature. This reduces joint mobility and strength and thus adversely affects amputees' ability to maintain balance. As a result, individuals with a LLA have been shown to fall more often when compared to age-matched and otherwise healthy individuals. In addition, individuals with LLA also have an increased fear of falling and reduced social participation because of this fear. Improving balance ability, reducing falls and fear of falling in this patient group through effective balance training interventions would have a number of socio-economic benefits. Such benefits may include but are not limited to reduced care costs, reduced burden on healthcare services and an improved sense of patient well-being. Therefore, the main aim of the current randomised control trial (RCT) is to investigate whether taking part in a games console based-balance intervention, improves experienced LLAs balance ability. The RCT also aims to assess how this intervention affects an amputee's falls rate, fear of falling and quality of life. After providing informed consent, unilateral lower limb amputees will be randomly allocated to one of two groups; an experimental group (12-week balance training intervention) or a control group (no intervention). Amputees in the experimental group will be loaned the use of a games console for the duration of the home-based intervention. Balance ability, falls rate, fear of falling and quality of life will be assessed prior to and post the intervention period as well as after three months following the end of the intervention period. Falls rate will also assessed one year post the intervention period. Results from the current study will provide evidence for the use of games-console based balance interventions in improving balance and falls outcomes for LLA.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputee to fit research design and must have at least 12 months experience using their prosthetic limb independently following discharge from in-patient treatment
* Minimum of 18 years old. There are no gender requirements - Age requirements in order to self-consent to participate, thus no child protection issues.
* Able to travel - Data collection takes place at University campus where participants will attend data collection sessions.
* Able to use prosthesis without pain or discomfort for a minimum of two hours at a time - Must be able to use prosthesis in order to complete tasks required for this research.
* Able to stand for periods of up to 2 minutes, unaided and without walking aid to complete tasks required for assessment where participants are required to stand on a force platform and perform some volitional postural movements.

Exclusion Criteria:

* Current musculoskeletal injury - Risk of further injury could be increased.
* Unable to follow instruction or cognitive deficits - Risk of further injury whilst completing tasks incorrectly.
* Bilateral amputation - In order to have a homogenous group of amputees in terms of categorisation of amputation.
* Unable to perform tasks due to current medical condition e.g. rheumatoid arthritis - Risk of worsening current condition and/or causing further injury.
* Experience pain or discomfort whilst wearing prosthesis - Risk of further injury and/or worsening of current condition. To be assessed by clinical team when individual is informed of study.
* Does not use prosthesis regularly.
* Not able to understand written and verbal English - All communication will be in English as the University does not have a service available that will be able to cope with translation demands.
* Currently taking medication known to affect balance adversely - Risk of falling during balance training and/or data collection sessions.
* Current Training - Participants must not be currently using the Nintendo Wii or similar systems in a structured balance training program.
* Inability to provide informed consent
* Substantial changes to the physical condition of the lower limb - If after consenting and participating in the study, individuals are referred to mobility services due to a degradation of the physical condition of either lower limb, they will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Limits of Stability Test Protocol Directional Control Score | Baseline to 3 Month Follow-Up
  Participants will also be required to complete the Limits of Stability test (LOS) which measures a participant's ability to perform postural movements in order to voluntarily move their centre of gravity (COG) as they stand on a force platform. The LOS requires participants to move their COG in the direction of eight pre-determined target directions as quickly and as accurately as possible. The eight pre-determined target directions will be representative of an individuals' 100% limit of stability based upon their height. Assuming that the body acts as an inverted pendulum with rotation about the ankle, this relates to the amount of movement possible before the COG position necessitates adjustment of the base of support by stepping. The directional control score (%) will be produced from this test protocol.
The Berg Balance Scale | Baseline to 3 Month Follow-Up
  Participants will complete the Berg Balance Scale, which involves the assessment of participants' ability to perform a number of functional tasks such as moving from standing to sitting, which are scored on a five point scale e.g. Needs assistance to sit (0) to sits safely with minimal use of hands (4). A total Berg Balance Scale score is calculated from this assessment.

SECONDARY OUTCOMES:
Falling | Baseline to 1 Year Follow-Up
  Falls, defined as an unexpected event in which the participant comes to rest on the ground, floor or lower level' will be recorded using prospective daily recording procedure with participants recording the occurrence of falls in a falls log book.
Falls Efficacy | Baseline to 3 Month Follow-Up
  Participants will complete the Modified Falls Efficacy scale in order to assess their falls efficacy.
The Prosthesis Evaluation Questionnaire | Baseline to 3 Month Follow-Up
  Participants will complete the Prosthesis Evaluation Questionnaire in order to assess their satisfaction with aspects concerning their prosthesis and their associated function.
The Short form-36 Questionnaire | Baseline to 3 Month Follow-Up
  Participants will complete the Short form-36 questionnaire to assess their quality of life.
The Activities and Balance Confidence Scale | Baseline to 3 Month Follow-Up
  Participants will complete the Activities and Balance Confidence Scale in order to assess their confidence in maintaining balance during activities of daily living.
Centre of Mass Dynamics | Baseline to 3 Month Follow-Up
  Participants biomechanical function, specifically the dynamics (movement) of their centre of mass, during the Limits of Stability Test protocol will be assessed in order to understanding the underpinning mechanisms of balance in this population.
Limits of Stability Test Protocol Maximal Excursion Score | Baseline to 3 Month Follow-Up
  Participants will also be required to complete the Limits of Stability test (LOS) which measures a participant's ability to perform postural movements in order to voluntarily move their centre of gravity (COG) as they stand on a force platform. The LOS requires participants to move their COG in the direction of eight pre-determined target directions as quickly and as accurately as possible. The eight pre-determined target directions will be representative of an individuals' 100% limit of stability based upon their height. Assuming that the body acts as an inverted pendulum with rotation about the ankle, this relates to the amount of movement possible before the COG position necessitates adjustment of the base of support by stepping. The maximal excursion score (%) will be produced from this test protocol.
Limits of Stability Test Protocol Reaction Time Score | Baseline to 3 Month Follow-Up
  Participants will also be required to complete the Limits of Stability test (LOS) which measures a participant's ability to perform postural movements in order to voluntarily move their centre of gravity (COG) as they stand on a force platform. The LOS requires participants to move their COG in the direction of eight pre-determined target directions as quickly and as accurately as possible. The eight pre-determined target directions will be representative of an individuals' 100% limit of stability based upon their height. Assuming that the body acts as an inverted pendulum with rotation about the ankle, this relates to the amount of movement possible before the COG position necessitates adjustment of the base of support by stepping. The reaction time score (s) will be produced from this test protocol.
Limits of Stability Test Protocol Movement Velocity Score | Baseline to 3 Month Follow-Up
  Participants will also be required to complete the Limits of Stability test (LOS) which measures a participant's ability to perform postural movements in order to voluntarily move their centre of gravity (COG) as they stand on a force platform. The LOS requires participants to move their COG in the direction of eight pre-determined target directions as quickly and as accurately as possible. The eight pre-determined target directions will be representative of an individuals' 100% limit of stability based upon their height. Assuming that the body acts as an inverted pendulum with rotation about the ankle, this relates to the amount of movement possible before the COG position necessitates adjustment of the base of support by stepping. The movement velocity score (degrees/second) will be produced from this test protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Cleveland T Barnett, Ph.D, Principal Investigator — Nottingham Trent University
Locations (2):
- United Kingdom (2):
  - The Biomechanics Lab, CELS Building, Nottingham Trent University, Nottingham, Notts
  - The Mobility Centre, City Hospital, NUH NHS Trust, Nottingham, Notts

IPD SHARING:
Plan to Share IPD: No